CLINICAL TRIAL: NCT04583865
Title: Assessment of the Feasibility and Quality of the Consultation by TeleConsultation in Pediatric Anesthesia in the Context of the Covid 19 Pandemic
Brief Title: Feasibility and Quality of TeleConsultation in Pediatric Anesthesia
Acronym: TéléCCCAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0220; 2020-A02275-34 (Registry Identifier: French ANSM register)
Record Dates: First submitted 2020-10-07; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia
Keywords: Teleconsultation-anesthesia
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- teleconsultation: Patient with teleconsultation of pre-anesthesia
  Interventions: Other: teleconsultation

INTERVENTIONS:
Other: teleconsultation — In the pandemic period linked to COVID, pediatric pre-anesthesis consultations should preferably be carried out by teleconsultation. This is to assess the effectiveness of these teleconsultation and the satisfaction of parents.

SUMMARY:
Teleconsultation (TLC) being a new method of anesthesia consultation, deployed as an emergency in healthcare facilities in the Covid context, it has never been evaluated either in terms of feasibility or in terms of quality. An initial assessment will highlight the pitfalls and difficulties encountered and suggest areas for improvement.

DETAILED DESCRIPTION:
The evaluation of teleconsultation in pediatric anesthesia, a new consultation method developed in the context of COVID for several weeks, appears necessary and will be a first inventory after its implementation in France. Analysis of the data collected in this study will allow us to propose technical, medical and organizational solutions to optimize the positioning and practical use of TLC for patients and care facilities. This assessment step seems imperative if the Covid context persists over time but could also be useful for the development of TLC outside the Covid context.

ELIGIBILITY:
Inclusion Criteria:

* All patients under the age of 18 requiring an anesthesia consultation for an act requiring anesthesia
* whose deprogramming in the context of the Covid 19 pandemic would lead to a loss of opportunity for the patient,
* Or whose programming in the context of the Covid 19 pandemic is in accordance with the recommendations made in field of the Professional Practice Recommendations
* And for which the family and the anesthetist have agreed to carry out the consultation by telemedicine

Exclusion Criteria:

* Patient whose anesthesia consultation is performed face-to-face as a first-line decision
* Family refusing teleconsultation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients under the age of 18 requiring an anesthesia consultation for an act requiring anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-09-14 (Estimated); Study Completion 2022-03-14 (Estimated)

PRIMARY OUTCOMES:
assess the feasibility of teleconsultation (TLC) in pediatric anesthesia in France in the context of the COVID 19 pandemic. | 3 months
  The feasibility of anesthesia TLC will be assessed by the failure rate of anesthesia TLC, defined by the conversion rate to degraded TLC (use of an unsecured video medium such as WhatsApp or simple audio communication without video support) or in face-to-face consultation

CONTACTS AND LOCATIONS:
Overall Officials: KERN Delphine, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No